CLINICAL TRIAL: NCT06383975
Title: Comparison Between VEin of MArshall Ethanol Infusion Versus Extended Pulmonary Vein PULSEd Field Ablation After Failed Pulmonary Vein Isolation in Patients with Persistent Atrial Fibrillation
Brief Title: VEin of MArshall Ethanolization Vs Extended Pulmonary Vein PULSEd Field Ablation After Failed PVI for Persistent AF
Acronym: VEMAPULSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sebastien Knecht (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Sebastien Knecht, Principal Investigator, AZ Sint-Jan AV
Organization: AZ Sint-Jan AV (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIV-24-01-045634
Record Dates: First submitted 2024-04-16; First posted 2024-04-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed field ablation with posterior wall isolation (Experimental)
  Interventions: Procedure: Pulsed field ablation with posterior wall isolation
- Radiofrequency ablation and vein of Marshall ethanolization (Active Comparator)
  Interventions: Procedure: Radiofrequency ablation and vein of Marshall ethanolization

INTERVENTIONS:
Procedure: Pulsed field ablation with posterior wall isolation — Extended pulmonary vein isolation including posterior wall isolation using pulsed field ablation
  Arms: Pulsed field ablation with posterior wall isolation
Procedure: Radiofrequency ablation and vein of Marshall ethanolization — Radiofrequency pulmonary vein re-isolation (when necessary), vein of Marshall ethanol infusion with roof and mitral lines
  Arms: Radiofrequency ablation and vein of Marshall ethanolization

SUMMARY:
The goal of this clinical trial is to compare two ablation techniques to treat patients with persistent atrial fibrillation (irregular and often very rapid heart rhythm). An ablation is a procedure during which some scars are made on the inside of the heart to break up the electrical signals that cause the irregular heartbeat. In this trial researchers will compare a new technique, which uses tiny electric shocks to make the scars, to the standard technique, which uses heat.

The main question the trial aims to answer is:

• Does the new technique work as well as the standard technique to prevent the irregular heartbeat from returning within one year of the procedure?

Participants will:

* Undergo an ablation with either the new or the standard technique
* Visit the hospital 1, 3, 6, 9 and 12 months after the procedure for a check-up
* Wear a device to register their heart rhythm for 24 hours before the 3 month visit and for 72 hours before the 6, 9 and 12 month visit
* Record their heart rhythm at home every week
* Complete a questionnaire 3, 6, 9 and 12 months after the procedure

DETAILED DESCRIPTION:
Background

Pulmonary vein isolation (PVI) remains the cornerstone of catheter ablation for the treatment of atrial fibrillation (AF). However, in patients with persistent AF, recurrence occurs in 20% to 50% of the patients. These patients often need additional ablation beyond PVI in the index procedure or in a redo procedure. During redo procedures, optimal management of AF has not been validated yet. Different strategies are used but without strong scientific background and without uniformity.

In the case of PV reconnection, PV re-isolation alone seems to be the gold standard in healthy atria, but with moderate success in patients with dilated left atrium or scar zones.

Different recent studies show a potential impact of posterior wall isolation; however with discordant results. This could be in part related to low rate of durable posterior wall isolation and also due to potential risk of esophageal fistula limiting the use of RF ablation at the posterior wall. The use of pulsed field energy could improve lesion durability and avoid any risk of fistula.

On the other hand, ethanol infusion in the vein of Marshal has also been shown to improve the success rate of persistent AF ablation but requires significant experience and may be time-consuming.

Rationale

Currently, there are no clear ablation endpoints in the case of AF recurrence post PVI. Especially for patients with persistent AF since substrate ablation beyond PVI does not seem to improve the success rate during a first procedure. However, this could be related to inappropriate patient selection. Indeed, PVI-resistant patients present those with worst prognosis with respect to AF recurrence. Additionally, when durable PVI is observed following recurrence in patients with persistent AF, case ablation beyond PVI seems reasonable and necessary.

The aim of this trial is to compare two strategies with clear endpoints, to avoid potential bias. The gold standard, PVI, is also respected in both groups In one group, PFA re-isolation of PVs and of the posterior wall has the advantage of a clear straight forward approach, with short-lasting procedures and which does not require high level technical skills.

In the second group, radiofrequency guided PV re-isolation will be performed in combination with mitral, aided by vein of Marshall ethanol infusion, and dome lines until bidirectional block. A Vein of Marshall is present in ~90% of the patients and strongly facilitates block at the mitral line (almost 100%) while a dome transection reduces the risk of further left atrial tachyarrhythmia.

Hypothesis

The hypothesis of this study is that the efficacy of a straightforward strategy of PV re-isolation (if necessary) and additional posterior wall isolation using the PFA FARAPULSETM catheter is comparable to that of a more complex and time consuming RF strategy aiming at vein of Marshall ethanol infusion and linear lesions at the roof and at the mitral line.

Design

This is a prospective, randomized (1:1), open label, blinded endpoint study (PROBE). Eligible subjects, who sign the study informed consent form, with persistent AF will be randomized into one of two study arms. In the pulsed field ablation (PFA) arm, patients will be treated using the FARAPULSETM catheter, aiming at pulmonary vein (PV) re-isolation (if necessary) and isolation of the posterior wall. In the radiofrequency (RF) group, patients will receive ethanol infusion in the vein of Marshall, followed by re-isolation of the PV (if necessary), dome and mitral lines with aim at bidirectional block.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent atrial fibrillation (AF) despite a first PVI. Persistent AF is defined as the presence of AF lasting ≥7 days (i.e. in case of new onset AF one has to wait for 7 days)

Exclusion Criteria:

* Persistent AF lasting ≥ 12 months
* Advanced valvular heart disease
* Left atrial (LA) volume >150mL
* LA diameter (PS-LAX) >60mm
* Septal wall diameter >15mm
* Life expectancy <1 year
* Weight >150 kg
* Any contra indication to catheter ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Atrial tachyarrhythmia recurrence within 12 months | 2-12 months
  Percentage of patients with any atrial tachyarrhythmia recurrence (> 30 sec) from 2 months (blanking period) to 12 months after the ablation procedure

SECONDARY OUTCOMES:
Safety and procedural related adverse event | During procedure-12 months
  Occurrence of vascular complications, tamponade, transient ischemic attack/stroke and other adverse events during and after the procedure, and within 12 months post procedure
Duration of the ablation procedure | During procedure
  Duration of the ablation procedure in both groups
Fluoroscopy time | During procedure
  Fluoroscopy time
Fluoroscopy dose | During procedure
  Fluoroscopy dose during the procedure
Effect of the procedure on quality of life | 3, 6, 9, 12 months
  Results of the 36-Item Short Form Survey Instrument (SF-36) before and 3, 6, 9 and 12 months post procedure. The scores range from 0 to 100. A higher score corresponds with a better outcome.
Incidence of repeat ablation | 12 months
  Percentage of patients who need another ablation within 12 months post procedure
Unscheduled visits and hospitalization | 12 months
  Number of unscheduled visits and hospitalization within 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Knecht, MD, PhD, Principal Investigator — AZ Sint-Jan Brugge AV
Locations (1):
- AZ Sint-Jan Brugge AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No